CLINICAL TRIAL: NCT04981977
Title: Examination of The Evidence-Based Care Transitions Intervention Enhanced With Peer Support to Reduce Racial Disparities in Hospital Readmissions and Negative Outcomes Post Hospitalization
Brief Title: Enhancing the Care Transitions Intervention With Peer Support to Reduce Disparities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Tampa General Hospital (Other); Lakeland Regional Health Medical Center (Unknown); AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY002687; AD-2019C1-16066 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Hospital Readmissions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Care Transitions Intervention (Experimental): Patient participants in this arm will receive the Care Transition Intervention.
  Interventions: Behavioral: Care Transitions Intervention
- Care Transition Intervention and Peer Support (Experimental): Patient participants in this arm will receive the Care Transition Intervention.
  Interventions: Behavioral: Care Transitions Intervention and Peer Support
- Usual Care (Other): Patient participants in this arm will receive the usual discharge/transition care provided by the hospital.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Care Transitions Intervention — CTI is delivered by a trained Care Transitions Coach (Coach) who works closely with patients to ensure a smooth transition from hospital to home following an acute hospitalization. The patient, caregiver, and Coach work together to maximize the involvement of interdisciplinary experts, ensuring that the appropriate professionals are involved, issues are addressed, goals are understood, and the discharge care plan is executed correctly. There are three aspects to CTI; the first is the initial hospital visit, followed by an in-home visit, concluding with telephone follow-up over a 28-day period. During these visits, the Coach focuses on four conceptual areas, referred to as pillars (i.e., Personal Health Record, Medication Management, Red Flags, and Physician Follow up). The Coach ensures the patient understands and utilizes the Personal Health Record to facilitate communication and ensure continuity of care plan across providers and settings.
  Other Names: CTI
  Arms: Care Transitions Intervention
Behavioral: Care Transitions Intervention and Peer Support — The PS intervention for this study is based upon the principles of motivational interviewing, which is a person-centered, goal-directed method to enhance intrinsic motivation for change by exploring and resolving ambivalence. A recent meta-analysis found the mean effect size for MI to be significantly larger for racial and ethnic minority samples (0.79 vs. 0.26) as compared to non-Hispanic Whites, highlighting its potential benefit and cultural relevance for minority populations. Patients in this arm of the study will receive the 28-day CTI intervention with a 2-month long Peer Support (PS) intervention provided by trained peer educators (PEs).
  Other Names: CTI + PS
  Arms: Care Transition Intervention and Peer Support
Other: Usual Care — The researchers will follow a control group of patients who meet study inclusion criteria. These older adults will participate in the traditional discharge case-management offered by the hospital where they were admitted and discharged. UC at our three partner hospitals consists of: (1) routine inpatient nurse intake that includes screening about housing, substance abuse, and functional status; (2) medication reconciliation performed by treating practitioners; (3) discharge patient education provided by inpatient nurses; (4) a list of resources for safety-net clinics and community-based services; and (5) for patients with severe chronic illness (e.g. heart failure) there may be a planned home visit by a nurse practitioner.
  Other Names: UC
  Arms: Usual Care

SUMMARY:
Unplanned hospital readmissions are extremely costly to patients and our healthcare system. Being readmitted to the hospital also leads to increased risk of health complications for patients including infections and impairments in functioning. Hospital readmissions are particularly common among older adults. Further, racial/ethnic disparities are evident in readmission rates and are the greatest among African American and Latino/Hispanic older adults. Effective, sustainable, and culturally appropriate interventions to improve outcomes, reduce unplanned hospital readmissions, and reduce health disparities are urgently needed. The proposed randomized controlled trial will evaluate the effectiveness of a novel transitional care strategy designed to avoid unplanned hospital readmissions and improve patient health outcomes in a racially/ethnically diverse sample of older adults who have been admitted to the hospital due to a chronic health condition.

Eric Coleman's Care Transitions Intervention (CTI) has been identified as the strategy most successfully implemented and evaluated in multiple settings and systems of care. CTI has been shown to reduce hospital readmissions for non-Hispanic White older adults, however its' effects have not been as strong for minority older adults in some studies and research trials have not recruited a sufficient number of racial/ethnic minorities to examine outcomes by race or ethnicity. Thus, it is unknown whether CTI is effective for racial/ethnic minority older adults who suffer disproportionately high readmission rates. Further, studies of transitions interventions suggest that older adult and racial/ethnic minority patients require additional assistance and support during transitions in care. The researchers hypothesize the addition of peer support will enhance and maximize the benefit of the CTI and increase its' cultural sensitivity and future sustainability.

The proposed 3-arm trial is designed to evaluate the Care Transitions Intervention (CTI) and CTI + Peer Support (PS), as compared to usual care (UC), on unplanned all-cause hospital readmissions occurring within 6 months (assessed at 30 days, 90 days and 6 months) and secondary health system (i.e., ED visits) and patient-centered outcomes (i.e., self-efficacy managing chronic disease, quality of life, functional status and mortality) among 402 hospitalized African American and Latino/Hispanic older adults (age 60+) who have a chronic physical illness (e.g., cardiovascular disease, diabetes, COPD) and are being discharged from the hospital back to the community.

DETAILED DESCRIPTION:
Unplanned hospital readmissions represent a critical failure of the healthcare system, perpetuate health disparities, and are the single largest driver of excess healthcare costs. For patients, hospital readmission increases risk for complications, infections, and functional impairment. Hospital readmissions are particularly prevalent among older adults. Further, racial/ethnic disparities in readmission rates are profound and are the greatest among African American and Latino/Hispanic older adults. Effective, sustainable and culturally appropriate interventions to improve outcomes, reduce un-planned hospital readmissions, and reduce health disparities are urgently needed. The proposed randomized controlled trial will evaluate the effectiveness of a novel transitional care strategy designed to avert un-planned hospital readmissions and improve patient health outcomes in a high-risk and under studied population of medically hospitalized African American and Latino/Hispanic older adults (age 60+). Transitional care strategies are interventions initiated before hospital discharge with the aim of ensuring the safe and effective transition of patients from the acute hospital setting to home. Of all the transitional care interventions tested, Eric Coleman's Care Transitions Intervention (CTI) has been identified as the strategy most successfully implemented and evaluated in multiple settings and systems of care. CTI is a non-clinical coaching strategy that occurs in the hospital, home, and via telephone for 28 days post-discharge.

CTI has been shown to reduce hospital readmissions for non-Hispanic White older adults, however intervention effects have been mixed for minority older adults and effectiveness trials have not recruited a sufficient number of racial/ethnic minorities to examine race or ethnicity specific outcomes. Thus, it is unclear whether CTI is effective for racial/ethnic minority older adults who suffer disproportionately high readmission rates. Further, studies of transitions interventions suggest that older adult and racial/ethnic minority patients require additional assistance and support during transitions in care. To address this gap, the researchers propose to add peer support (PS) to the CTI to enhance its effectiveness among high-risk populations of racial/ethnic minority older adults. The researchers believe the addition of peer support will enhance and maximize the benefit of the CTI and increase its' cultural sensitivity and future sustainability. The proposed 3-arm trial is designed to evaluate the Care Transitions Intervention (CTI) and CTI + Peer Support (PS), as compared to usual care (UC), on all cause unplanned hospital readmissions occurring within 6 months (assessed at 30 days, 90 days and 6 months) and secondary health system (i.e., ED visits) and patient-centered outcomes (i.e., self-efficacy managing chronic disease, quality of life, functional status and mortality) among 402 hospitalized African American and Latino/Hispanic older adults (age 60+) who have a chronic physical illness (e.g., cardiovascular disease, diabetes, COPD) and are being discharged from the hospital back to the community. The researchers will also maximize the uniquely diverse sample to explore potential mediators and moderators of intervention effects. The researchers will further conduct semi-structured interviews with patients (n=48) and caregivers (n=24) to qualitatively examine mechanisms impacting readmission risk and patient-centered outcomes post discharge. The researchers will utilize multi-methods to triangulate and contextualize the findings.

ELIGIBILITY:
Inclusion Criteria:

Patient participants (N=402) will be included in the study if they:

* Are aged 60+
* Identify as African American or Latino/Hispanic (any race)
* Are being discharged from one of our three hospital partners to home with no planned readmissions
* Have access to a household telephone or cellphone
* Speak English or Spanish

Exclusion Criteria:

Patient participants will be excluded from the study if they:

* Are younger than age 60
* Identify as any race/ethnicity other than African American or Latino/Hispanic
* Are being discharged with a condition that has planned readmission (e.g. transplant patient, chemotherapy etc.)
* Are permanent residents of a skilled nursing facility, receiving hospice service, or are being discharged to a long-term care facility
* Have a comorbid substance use disorder
* Are actively suicidal or homicidal
* Have a comorbid psychotic disorder or organic mental disorder (e.g., dementia)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Unplanned All-Cause Hospital Readmissions | 30 days
  The researchers will evaluate the Care Transitions Intervention (CTI) and CTI + Peer Support (PS), compared to usual care (UC), on the primary outcome of unplanned all-cause hospital readmissions using data from the Florida Health Information Exchange (HIE) Services Electronic Notification System (ENS).
Unplanned All-Cause Hospital Readmissions | Three months
  The researchers will evaluate the Care Transitions Intervention (CTI) and CTI + Peer Support (PS), compared to usual care (UC), on the primary outcome of unplanned all-cause hospital readmissions using data from the Florida Health Information Exchange (HI
Unplanned All-Cause Hospital Readmissions | Six months
  The researchers will evaluate the Care Transitions Intervention (CTI) and CTI + Peer Support (PS), compared to usual care (UC), on the primary outcome of unplanned all-cause hospital readmissions using data from the Florida Health Information Exchange (HI
Related Secondary Health-System Visits (i.e., ED Visits) | 30 days
  The researchers will evaluate the Care Transitions Intervention (CTI) and CTI + Peer Support (PS), compared to usual care (UC), on the primary outcome of unplanned related secondary health-system visits using data from the Florida Health Information Exchange (HIE) Services Electronic Notification System (ENS).
Related Secondary Health-System Visits (i.e., ED Visits) | Three months
  The researchers will evaluate the Care Transitions Intervention (CTI) and CTI + Peer Support (PS), compared to usual care (UC), on the primary outcome of unplanned related secondary health-system visits using data from the Florida Health Information Exchange (HIE) Services Electronic Notification System (ENS).
Related Secondary Health-System Visits (i.e., ED Visits) | Six months
  The researchers will evaluate the Care Transitions Intervention (CTI) and CTI + Peer Support (PS), compared to usual care (UC), on the primary outcome of unplanned related secondary health-system visits using data from the Florida Health Information Exchange (HIE) Services Electronic Notification System (ENS).

SECONDARY OUTCOMES:
Demographic Questionnaire | At time of enrollment/Baseline
  All participants be asked a series of demographic questions, which include self-reported: race, ethnicity, gender, education, employment status, health insurance status, immigration status marital status, exposure to violence, number of children, and self-rated health.
Care Transitions Measure (CTM-3) | 30 days
  The Care Transitions Measure (CTM-3) assesses the extent to which essential care was performed by hospital staff when planning to discharge a patient from the hospital and engage them in posthospital self-care activities (Antchkova et al., 2014). The 3-item CTM accounts for 88% of variance in the original 15-item CTM score (Parry et al., 2008).
Care Transitions Measure (CTM-3) | Three months
  The Care Transitions Measure (CTM-3) assesses the extent to which essential care was performed by hospital staff when planning to discharge a patient from the hospital and engage them in posthospital self-care activities (Antchkova et al., 2014). The 3-item CTM accounts for 88% of variance in the original 15-item CTM score (Parry et al., 2008).
Care Transitions Measure (CTM-3) | Six months
  The Care Transitions Measure (CTM-3) assesses the extent to which essential care was performed by hospital staff when planning to discharge a patient from the hospital and engage them in posthospital self-care activities (Antchkova et al., 2014). The 3-item CTM accounts for 88% of variance in the original 15-item CTM score (Parry et al., 2008).
Self-Efficacy (SES-6) | Baseline
  The SES-6 is a 6-item scale that was developed for the Chronic Disease Self-Management Study that assess for emotional functioning, role function, symptom control, and communication with physicians (Lorig et al., 2001).
Self-Efficacy (SES-6) | 30
  The SES-6 is a 6-item scale that was developed for the Chronic Disease Self-Management Study that assess for emotional functioning, role function, symptom control, and communication with physicians (Lorig et al., 2001).
Self-Efficacy (SES-6) | Three months
  The SES-6 is a 6-item scale that was developed for the Chronic Disease Self-Management Study that assess for emotional functioning, role function, symptom control, and communication with physicians (Lorig et al., 2001).
Self-Efficacy (SES-6) | Six months
  The SES-6 is a 6-item scale that was developed for the Chronic Disease Self-Management Study that assess for emotional functioning, role function, symptom control, and communication with physicians (Lorig et al., 2001).
Medical Outcomes Study Short Form (MOS SF-36) | Baseline
  The RAND MOS SF-36 was adapted from the SF-36 for use in an observational study that measured differences in the practicing styles of physicians and patient outcomes. It assesses for 8 health concepts: (1) physical functioning; (2) bodily pain; (3) limitations in physical activity due to health challenges; (4) limitations in social activities due to due to physical or emotional challenges; (5) general health perceptions; (6) energy and fatigue (vitality); (7) emotional well-being; and (8) social functioning (Ware & Sherbourne, 1992).
Medical Outcomes Study Short Form (MOS SF-36) | 30 days
  The RAND MOS SF-36 was adapted from the SF-36 for use in an observational study that measured differences in the practicing styles of physicians and patient outcomes. It assesses for 8 health concepts: (1) physical functioning; (2) bodily pain; (3) limitations in physical activity due to health challenges; (4) limitations in social activities due to due to physical or emotional challenges; (5) general health perceptions; (6) energy and fatigue (vitality); (7) emotional well-being; and (8) social functioning (Ware & Sherbourne, 1992).
Medical Outcomes Study Short Form (MOS SF-36) | Three months
  The RAND MOS SF-36 was adapted from the SF-36 for use in an observational study that measured differences in the practicing styles of physicians and patient outcomes. It assesses for 8 health concepts: (1) physical functioning; (2) bodily pain; (3) limitations in physical activity due to health challenges; (4) limitations in social activities due to due to physical or emotional challenges; (5) general health perceptions; (6) energy and fatigue (vitality); (7) emotional well-being; and (8) social functioning (Ware & Sherbourne, 1992).
Medical Outcomes Study Short Form (MOS SF-36) | Six months
  The RAND MOS SF-36 was adapted from the SF-36 for use in an observational study that measured differences in the practicing styles of physicians and patient outcomes. It assesses for 8 health concepts: (1) physical functioning; (2) bodily pain; (3) limitations in physical activity due to health challenges; (4) limitations in social activities due to due to physical or emotional challenges; (5) general health perceptions; (6) energy and fatigue (vitality); (7) emotional well-being; and (8) social functioning (Ware & Sherbourne, 1992).
Quality of Life (WHOQOL-BRIEF) | Baseline
  The WHOQOL-BREF is a 26-item self-report questionnaire that addresses 4 QOL domains: (1) social relationships (3 items); (2) psychological health (6 items); (3) physical health (7 items); and (4) environment (8 items). Two other general health and QOL items are also included.
Quality of Life (WHOQOL-BRIEF) | 30 days
  The WHOQOL-BREF is a 26-item self-report questionnaire that addresses 4 QOL domains: (1) social relationships (3 items); (2) psychological health (6 items); (3) physical health (7 items); and (4) environment (8 items). Two other general health and QOL items are also included.
Quality of Life (WHOQOL-BRIEF) | Three months
  The WHOQOL-BREF is a 26-item self-report questionnaire that addresses 4 QOL domains: (1) social relationships (3 items); (2) psychological health (6 items); (3) physical health (7 items); and (4) environment (8 items). Two other general health and QOL items are also included.
Quality of Life (WHOQOL-BRIEF) | Six months
  The WHOQOL-BREF is a 26-item self-report questionnaire that addresses 4 QOL domains: (1) social relationships (3 items); (2) psychological health (6 items); (3) physical health (7 items); and (4) environment (8 items). Two other general health and QOL items are also included.
Medication Management (MedMaleDE) | Baseline
  The Medication Management Instrument for Deficiencies in the Elderly (MedMalDE), assesses for three domains: (1) what the person knows about their medications; (2) whether a person knows how to take their medications; and (3) whether the person knows how to get their medications.
Medication Management (MedMaleDE) | 30 days
  The Medication Management Instrument for Deficiencies in the Elderly (MedMalDE), assesses for three domains: (1) what the person knows about their medications; (2) whether a person knows how to take their medications; and (3) whether the person knows how to get their medications.
Medication Management (MedMaleDE) | Three months
  The Medication Management Instrument for Deficiencies in the Elderly (MedMalDE), assesses for three domains: (1) what the person knows about their medications; (2) whether a person knows how to take their medications; and (3) whether the person knows how to get their medications.
Medication Management (MedMaleDE) | Six months
  The Medication Management Instrument for Deficiencies in the Elderly (MedMalDE), assesses for three domains: (1) what the person knows about their medications; (2) whether a person knows how to take their medications; and (3) whether the person knows how to get their medications.
Satisfaction Survey | Six months
  Patient participants will complete a brief satisfaction survey at their last follow-up assessment to learn more about their experience participating in this research project and to learn about why they chose to participate in this research project.
Caregiver Qualitative Interview | Six months
  A random selection of patient participants will participate in a one-hour interview with a study GRA at the end of the project. The focus of the interview is to learn more about their experience participating in this project, and to get their perspective on how it has benefited/or not benefited them.

CONTACTS AND LOCATIONS:
Overall Officials: Amber M Gum, Phd, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided